CLINICAL TRIAL: NCT01148784
Title: A Prospective Randomized Comparison of Doubled Versus Quadrupled Allogenic Tissue Constructs for Anterior Cruciate Ligament Reconstruction
Brief Title: Comparison of Doubled Quadrupled Versus Quadrupled Allograft Tissue Constructs for Anterior Cruciate Ligament (ACL) Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Dennis Crawford, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OHSU-6158
Record Dates: First submitted 2010-06-21; First posted 2010-06-22 (Estimated); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Anterior Cruciate Ligament; Injury
Keywords: anterior cruciate ligament tear; ACL; ligament; knee; allograft
MeSH Terms: conditions — Wounds and Injuries; Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quadrupled Hamstring Allograft (Active Comparator)
  Interventions: Procedure: ACL reconstruction
- Doubled Tibialis Anterior Allograft (Active Comparator)
  Interventions: Procedure: ACL reconstruction

INTERVENTIONS:
Procedure: ACL reconstruction — Randomized comparison of two different allogenic tissue types, quadrupled hamstring or doubled tibialis anterior, for anterior cruciate ligament repair.

SUMMARY:
The purpose of this study is to compare two different soft tissue allografts, double bundle tibialis anterior allograft or quadruple bundle hamstring allograft, used in repairing a torn anterior cruciate ligament (ACL) of the knee.

ELIGIBILITY:
Inclusion Criteria:

* ACL injury is the primary limitation to activities of daily living.

Exclusion Criteria:

* Multiple current ligamentous injuries to the knee.
* Revision reconstruction of the ACL.
* Uncorrected instability of the ACL on the opposite knee.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2010-06; Primary Completion 2012-09-17 (Actual); Study Completion 2014-04-05 (Actual)

PRIMARY OUTCOMES:
Knee outcome scores | One year
  The change of physical function and pain as evaluated by patient reported outcome measures (Knee injury and Osteoarthritis Outcome Score (KOOS), International Knee Documentation Committee (IKDC) score).

CONTACTS AND LOCATIONS:
Overall Officials: Dennis C Crawford, MD, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States